CLINICAL TRIAL: NCT04074174
Title: Investigation of the Effect of NNC0174-0833 on Pharmacokinetics of an Oral Combination Contraceptive (Ethinylestradiol and Levonorgestrel) in Females of Non-childbearing Potential
Brief Title: Research Study to Investigate the Effect of NNC0174-0833 on a Birth Control Pill in Women Who Are Not Able to Become Pregnant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-4517; U1111-1228-4219 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Contraceptives, Oral; Tablets; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NNC0174-0833 treatment-free period; NNC0174-0833 treatment (Experimental): During the NNC0174-0833 treatment-free period participants will receive OC tablets and acetaminophen. During the NNC0174-0833 treatment period participants will receive OC tablets and acetaminophen in addition to NNC0174-0833.
  Interventions: Drug: NNC0174-0833; Drug: Oral contraceptive (OC) tablets; Drug: Acetaminophen

INTERVENTIONS:
Drug: NNC0174-0833 — NNC0174-0833 administered s.c. (subcutaneously, under the skin) once weekly for 12 weeks
Drug: Oral contraceptive (OC) tablets — 1 tablet daily on days 1-8 and days 79-86
Drug: Acetaminophen — Single dose of acetaminophen as part of a standardised meal on day 1 and day 79

SUMMARY:
The study looks at how the study medicine affects the level in the blood of a birth control pill. The study also looks at how the study medicine affects the duration of emptying of the stomach. Participants will get 1 injection of study medicine once a week for 12 weeks by a study nurse at the clinic. The study medicine is injected with a thin needle in a skin fold in the stomach. In addition, participants will get 1 birth control pill per day for 8 days before the first dose of the study medicine and again after 10 weeks of dosing with the study medicine. Participants will also get a dose of acetaminophen before the first dose of the study medicine and again after 10 weeks of dosing with the study medicine. Acetaminophen is a mild painkiller but used here to assess the emptying of the stomach. The study will last for about 9 months, but participants will only be in the study for about 6 months. Participants will have 17 clinic visits with the study staff and some will be overnight visits. There will also be 3 phone calls with the study staff. At all visits, participants will have blood drawn along with other clinical assessments. Participants will be asked about their health, diseases and habits including mental health questionnaires. Participants must not be able to become pregnant if they want to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential, aged 18-65 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 25.0 and 39.9 kg/m^2 (both inclusive). Overweight should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products (including acetaminophen) or related products.
* Previous participation in this trial. Participation is defined as signed informed consent.
* Previous participation in trial(s) with NNC0174-0833 unless documented that the subject was assigned to placebo treatment. Participation is defined as randomised.
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,EE,SS area under the ethinylestradiol concentration-time curve during a dosing interval (0-24 hours) at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  h*pg/mL
AUC0-24h,LN,SS area under the levonorgestrel concentration-time curve during a dosing interval (0-24 hours) at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  h*pg/mL

SECONDARY OUTCOMES:
Cmax,EE, SS, maximum concentration of ethinylestradiol at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  pg/mL
Cmax,LN,SS, maximum concentration of levonorgestrel at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  pg/mL
tmax,EE,SS time to maximum concentration of ethinylestradiol at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  h
tmax,LN,SS, time to maximum concentration of levonorgestrel at steady state | Day 8 (predose to 24 hours post-dose) and Day 79 (predose to 24 hours post-dose)
  h
AUC0-60min,para, area under the acetaminophen (paracetamol) concentration-time curve for 0-60 minutes following a standardised meal | Day 1 (predose to 60 minutes post-dose) and Day 79 (predose to 60 minutes post-dose)
  h*microg/mL
AUC0-360min,para, area under the acetaminophen (paracetamol) concentration-time curve for 0-360 minutes following a standardised meal | Day 1 (predose to 360 minutes post-dose) and Day 79 (predose to 360 minutes post-dose)
  h*microg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com